CLINICAL TRIAL: NCT06133101
Title: Impact of Soymilk on Liver Disease Severity of Children With Non-alcoholic Fatty Liver Disease (NAFLD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Marialena Mouzaki (Other)
Responsible Party: Sponsor-Investigator, Marialena Mouzaki, Professor, Division of Gastroenterology, Hepatology and Nutrition, Children's Hospital Medical Center, Cincinnati
Organization: Children's Hospital Medical Center, Cincinnati (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0416
Record Dates: First submitted 2023-10-13; First posted 2023-11-15 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Prospective parallel arm randomized controlled study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 2% Fat Cows Milk (Placebo Comparator): Participants randomized to this arm will consume 2% fat cow's milk twice daily for 12 weeks.
  Interventions: Drug: 2% Fat Cow's Milk
- Standard Soy Milk (Experimental): Participants randomized to this arm will consume standard soy milk twice daily for 12 weeks.
  Interventions: Drug: Standard Soy Milk

INTERVENTIONS:
Drug: Standard Soy Milk — Consumption of commercially available soy milk
  Arms: Standard Soy Milk
Drug: 2% Fat Cow's Milk — Consumption of commercially available 2% cow's milk
  Arms: 2% Fat Cows Milk

SUMMARY:
A randomized, controlled study of standard soy milk consumption compared to 2% fat cow's milk consumption in children with Non-alcoholic Fatty Liver Disease (NAFLD). The investigators hypothesize that the daily consumption of soy isoflavones found in the soy milk will be beneficial in reducing NAFLD and other obesity-related comorbidities. The investigators do not expect any adverse endocrine or metabolomic effects from the consumption of soy isoflavones.

ELIGIBILITY:
Inclusion Criteria:

* Children with overweight/obesity
* Non-alcoholic fatty liver disease (NAFLD) and an MRI PDFF >10%
* Known NAFLD or elevated ALT for sex (>22 for females and >26 for males)

Exclusion Criteria:

* MRI-PDFF <10%
* Baseline habitual (>3 days per week) consumption of soy foods
* Allergy to soy or cow's milk protein
* Inability to undergo MRI
* Recent (past 8 weeks) antibiotic exposure
* Treatment for existing endocrine disorders

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in liver disease severity | 12 weeks
  Change in liver disease severity, measured using magnetic resonance imaging-proton density fat fraction (MRI-PDFF). A relative PDFF change of 30% correlates with histologic improvement in patients with NAFLD and is commonly used in clinical trials.

SECONDARY OUTCOMES:
Change in serum aminotransferase levels (ALT, aspartate aminotransferase [AST], GGT, alkaline phosphatase [ALP]) | 12 weeks
Change in gamma glutamyl-transferase levels (GGT) | 12 weeks
Change in alkaline phosphatase (ALP) | 12 weeks
Change in fasting triglycerides | 12 weeks
Change in total cholesterol (TC) | 12 weeks
Change in high- and low-density lipoprotein (HDL-C, LCL-C) levels | 12 weeks
Change in glucose | 12 weeks
Change in insulin | 12 weeks
Change in glycated hemoglobin (HbA1c) | 12 weeks
Change in testosterone, estrogen and sex hormone binding globulin (SHBG) levels | 12 weeks
Change in thyroid function (TSH and Free T4) | 12 weeks
Change in estradiol | 12 weeks
Change in serum metabolome and lipidome | 12 weeks
Change in systolic and diastolic blood pressure | 12 weeks
Change in equol production status | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States